CLINICAL TRIAL: NCT01012596
Title: Effectiveness, Intention, and Behavior in Creighton Model NFP Use
Brief Title: Creighton Model Effectiveness, Intentions and Behaviors Assessment (CEIBA)
Acronym: CEIBA
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Joseph B. Stanford, MD, MSPH, Principal Investigator, University of Utah
Other Study IDs: 34487; PA-FPR-08-38; PA-FPR-001-009858; CEIBA-93.974
Record Dates: First submitted 2009-11-02; First posted 2009-11-13 (Estimated); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Pregnancy; Fertility
Keywords: Natural Family Planning Methods; Ovulation Detection; Cervix Mucus; Intention; Behavior; Birth Control; Contraception; Pregnancy; Fertility
MeSH Terms: conditions — Behavior | interventions — Natural Family Planning Methods; Ovulation Detection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Creighton Model: New and return users of the Creighton Model FertilityCare System, a method of Natural Family Planning.
  Interventions: Behavioral: Creighton Model System of Natural Family Planning

INTERVENTIONS:
Behavioral: Creighton Model System of Natural Family Planning — Participants will learn the Creighton Model, a standardized method of natural family planning, from FertilityCare Practitioners from established FertilityCare Centers. The learning can be done in-person or long distance.
  Other Names: Natural Family Planning; Ovulation Method; Fertility Awareness

SUMMARY:
The Creighton Model (CrM) FertilityCare System is a natural family planning method that teaches couples to recognize and chart the signs of fertility and infertility in the woman's cycle and to use that knowledge to either achieve or avoid a pregnancy. The method is natural, safe and effective, and it helps the couple understand their fertility. Trained practitioners at FertilityCare Centers teach the Creighton Model across the country, internationally and long distance.

Several FertilityCare Centers and the University of Utah are conducting a study to evaluate the effectiveness of the Creighton Model (CrM) for new and return users wanting to avoid pregnancy. While past studies have shown that the Creighton Model is a highly effective method, this study will use new ways to measure how well it works. This is important because the knowledge gained will improve comparisons between the Creighton Model and other family planning methods. The study will also explore intentions and behaviors of couples to avoid or achieve a pregnancy.

The investigators hypothesize that for the CrM the pregnancy rate during perfect use to avoid pregnancy will be about 1% and the behaviorally determined avoiding-related pregnancy rate for the CrM will be about 6%. The investigators will also evaluate the pregnancy rate during "typical use" without a previously stated intention to conceive (in CrM terms, a mixture of avoiding and achieving-related behavior).

DETAILED DESCRIPTION:
There are a variety of natural family planning (NFP) methods available today that differ in algorithm and biomarkers used to identify women's fertile window. This study will directly evaluate the NFP system known as the Creighton Model FertilityCare System (CrM). The Creighton Model System is a well-established educational system about fertility which involves no devices. The CrM teaches women a standardized way of observing and describing their vaginal discharge each day during routine use of the bathroom, and interpreting the changes in vaginal discharge to determine whether they are likely to be fertile that day or not. Vaginal discharge changes as tracked by the CrM are an accurate indicator of the changes in secretions from the uterine cervix that relate to the approach of ovulation.

This study will also examine the relationship between a couple's stated intentions to achieve or avoid a pregnancy during each menstrual cycle with their sexual behavior during the same cycle. There is growing consensus among researchers that current measures of pregnancy intention are simplistic at best, and at worst can be very misleading. One of the purposes of the study is to explore the multiple dimensions of pregnancy motivations, intentions, and behaviors by newer detailed measures.

This study will enroll couples who are new or returning CrM users and who are trying to avoid a pregnancy at the time they begin use of the CrM. The participants will be recruited from CrM FertilityCare Centers. The design is a prospective cohort study, which is the optimal study design to assess different measures of effectiveness and intendedness simultaneously in a group of NFP users. Several of the key measures of intention and behavior required for this study must be assessed prior to the outcome of actual use of CrM over time and the outcome of pregnancy, to avoid recall bias. Outcomes for this study require relatively precise assessment of the timing of both intentions and behaviors, which is simply unavailable from recall. We plan to enroll at least 300 and up to 400 couples in the study. This represents 60% (300/497) of the estimated available and eligible couples learning the CrM for use to avoid pregnancy in one year at the participating FertilityCare Centers.

ELIGIBILITY:
Inclusion Criteria:

* Being a new or return user of the Creighton Model with the stated intention of avoiding pregnancy
* Sexually active or planning to be sexually active within 6 months of the enrollment date (relevant to some engaged couples who learn CrM)
* The woman is between the ages of 18 to 40
* The man is age 18 or older
* The woman has had at least 2 menstrual flows in the past 3 months or at least one menstrual flow since stopping hormonal birth control
* The woman is able to complete questionnaires in English

Exclusion Criteria:

* History of infertility
* Confirmed pelvic inflammatory disease, surgically confirmed untreated endometriosis, chemotherapy (either man or woman), or radiation to the reproductive tract (either man or woman)
* Hysterectomy, oophorectomy (ovary removed), tubal ligation, fallopian tube surgery, surgery for ectopic pregnancy, removal of a testicle (orchiectomy) or vasectomy
* Depo-Provera injection any time in the past 2 years
* Totally breastfeeding an infant, without any supplements

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will enroll couples who are new or return Creighton Model (CrM) users and who are trying to avoid a pregnancy at the time they begin use of the CrM. The participants will be recruited from several CrM FertilityCare Centers across the United States and Canada. Participants who do not live near a center will be offered long distance teaching.
Sampling Method: Non-Probability Sample
Enrollment: 624 (Actual)
Dates: Start 2009-10; Primary Completion 2012-10 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Pregnancy rates during perfect and typical use of the Creighton Model FertilityCare System (CrM) to avoid pregnancy in a way directly comparable to the approach used in recent family planning effectiveness studies | 1 year

SECONDARY OUTCOMES:
The intention status of all pregnancies according to standard measures of intended, mistimed and unwanted pregnancy while recognizing the significant limitations of these measures | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B Stanford, MD, MSPH, Principal Investigator — University of Utah
Locations (18):
- United States (17):
  - Sacramento Diocese FertilityCare Services, Sacramento, California
  - Northland Family Programs: A FertilityCare Center, Duluth, Minnesota
  - Twin Cities FertilityCare Center, Saint Paul, Minnesota
  - FertilityCare Center of Kansas City, Blue Springs, Missouri
  - St. John's Mercy Medical Center, Department of FertilityCare Services, St Louis, Missouri
  - FertilityCare Center, Diocese of Lincoln, Lincoln, Nebraska
  - FertilityCare Center of Omaha, Omaha, Nebraska
  - FertilityCare Services St. Joseph Hospital, Nashua, New Hampshire
  - St. Joseph FertilityCare Center, Albuquerque, New Mexico
  - Caritas FertilityCare Center, Pataskala, Ohio
  - Center for Women's Health, Spirit FertilityCare Services, Camp Hill, Pennsylvania
  - FertilityCare Services: Diocese of Charleston, SC, Greer, South Carolina
  - FertilityCare Center of North Texas, Fort Worth, Texas
  - Women's FertilityCare Services of Houston, Houston, Texas
  - Intermountain FertilityCare Center, Salt Lake City, Utah
  - If you don't find a center near you, contact us for Long Distance Learning, Salt Lake City, Utah
  - FertilityCare Center of the Upper Ohio Valley, Weirton, West Virginia
- Marguerite Bourgeoys FertilityCare Programme, Toronto, Ontario, Canada

REFERENCES:
- See also: Study Website — https://medicine.utah.edu/dfpm/public-health/research/ocrh/studies/ceiba.php